CLINICAL TRIAL: NCT06111846
Title: An Open-label Phase IIa Study to Evaluate the Safety and Preliminary Efficacy of HBMMSC Injection in the Treatment of APAP
Brief Title: Study of Human Bone Marrow Mesenchymal Stem Cells in APAP
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiuzhitang Maker (Beijing) Cell Technology Co.,Ltd. (Other)
Collaborators: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MKMSC-CT-001
Record Dates: First submitted 2023-10-19; First posted 2023-11-01 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Autoimmune Pulmonary Alveolar Proteinosis
MeSH Terms: conditions — Pulmonary Alveolar Proteinosis, Acquired

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: hBMMSC (Experimental): 1.0×10^6/kg hBMMSC (participant's body weight) single dose 2.0×10^6/kg hBMMSC (participant's body weight) single dose 2.0×10^6/kg hBMMSC (participant's body weight) administered twice
  Interventions: Drug: human Bone Marrow Mesenchymal Stem Cell (hBMMSC)

INTERVENTIONS:
Drug: human Bone Marrow Mesenchymal Stem Cell (hBMMSC) — Group 1: 1.0×10^6 cells/kg (participant's body weight) single dose (n=3) Group 2: 2.0×10^6 cells/kg (participant's body weight) single dose (n=3) Group 3: 2.0×10^6 cells/kg (participant's body weight) administered twice (n=4)
  Other Names: hBMMSC

SUMMARY:
The purpose of this open-label phase IIa clinical trial study is to evaluate the safety and preliminary efficacy of hBMMSC intravenous treatment in patients with aPAP.

DETAILED DESCRIPTION:
Autoimmune pulmonary alveolar proteinosis (aPAP) is a rare lung disease for which there is no specific drug treatment. Currently, the standard treatment strategy for PAP is whole-lung lavage (WLL), which is invasive and has limited therapeutic efficacy. The purpose of this study is to evaluate the safety and preliminary efficacy of hBMMSC intravenous treatment in patients with aPAP. The clinical trial intends to involve 10 participants. The trial is expected to last approximately 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or older
* Patients diagnosed with aPAP by both CT and biopsy (TBLB, TBCB, or surgical lung biopsy) or bronchoalveolar perfusion (BAL) as well as GM-CSF autoantibodies in serum positive
* No remission was demonstrated by CT, pulmonary function test results,or blood gas analysis at least 2 times (at least 3 months apart) before enrollment
* At rest PaO2≤70 mmHg
* Fertile participants must receive effective medical contraception (for both male and female participants, up to one year after the last study dosing)
* Voluntary signed informed consent

Exclusion Criteria:

* Diagnosed with hereditary PAP, secondary PAP, or another type of PAP
* Received whole lung lavage（WLL） therapy within 6 months before enrollment
* Received previous GM-CSF therapy within 6 months before enrollment
* Received other clinical trial treatment within 3 months before enrollment
* Participated in other stem cell studies within 1 year before enrollment
* Inflammatory disease or autoimmune disorder requiring treatment associated with significant immunosuppression (e.g. more than 10 mg/day systemic prednisolone)
* Active infection (viral, bacterial, fungal or mycobacterial), which may affect the assessment of efficacy in the trial
* History of malignant tumors
* Known allergic reactions to any of the ingredients in the study drug
* Participants who, in the opinion of the investigator, would aggravate any other serious pre-existing medical condition are not suitable for this trial
* Women who are known to be pregnant, breastfeeding, have a positive pregnancy test (which will be detected during the screening process), or plan to become pregnant during the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-12-25 (Actual); Primary Completion 2025-07-22 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Alveolar-arterial difference in oxygen tension (A-aDO2) | 24 weeks
  The changes of alveolar-arterial difference in oxygen tension (A-aDO2) relative to baseline were assessed in the hBMMSC treated group after 24 weeks of treatment.

SECONDARY OUTCOMES:
Safety and tolerability | 48 weeks
  Number of participants with serious and non-serious adverse events
Difference in pulmonary function | 4 weeks, 12 weeks, 24 weeks, 48 weeks
  Pulmonary function tests include diffusing capacity of the lung for carbon monoxide(DLCO),forced vital capacity(FVC), forced expiratory volume in one second(FEV1).Change from Baseline in the DLCO、FVC、 FEV1 as measured
Alveolar-arterial oxygen difference (A-aDO2) | 48 weeks
  Change from Baseline in the A-aDO2 as measured
Difference in 6-minute walk distance (6MWD) | 4 weeks, 12 weeks, 24 weeks, 48 weeks
  Change from Baseline in the 6MWD as measured
Percutaneous arterial oxygen saturation (SpO2) | 4 weeks, 12 weeks, 24 weeks, 48 weeks
  Change from Baseline in the SpO2 as measured
Difference in modified Medical Research Council（mMRC） | 4 weeks, 12 weeks, 24 weeks, 48 weeks
  Change from Baseline in the mMRC as tested
Difference in St. George's Respiratory Questionnaire（SGRQ） | 4 weeks, 12 weeks, 24 weeks, 48 weeks
  Change from Baseline in the SGRQ as tested
Imaging（Chest CT score ） | 24 weeks, 48 weeks
  Parenchymal lung density determined by quantitative computed tomography (CT) densitometry. Change from Baseline (Day 0) in the parenchymal densitometry as measured at 24 and 48 weeks
Difference in Disease severity score (DSS) | 24 weeks, 48 weeks
  Change from Baseline in the DSS score
Difference in arterial partial pressure of oxygen (PaO2) | 24 weeks, 48 weeks
  Change from Baseline in the PaO2 as measured
Difference in Krebs Von den Lungen-6（KL-6） | 2 weeks，4 weeks, 12 weeks, 24 weeks
  Change from Baseline in the KL-6 as measured
Difference in carcinoembryonic antigen（CEA） | 2 weeks，4 weeks, 12 weeks, 24 weeks
  Change from Baseline in the CEA as measured
Difference in lactate dehydrogenase (LDH) | 2 weeks，4 weeks, 12 weeks, 24 weeks
  Change from Baseline in the LDH as measured
Number of Rescue whole lung lavage (WLL) in 108 weeks | 108 weeks
  Criteria for performing WLL were based on symptoms, decreased exercise capacity, and/or worsening of clinical symptoms of aPAP as judged by the investigator that the participant developed hypoxemia or decreased oxygen saturation

CONTACTS AND LOCATIONS:
Locations (1):
- JiuzhitangMakerBeijingCellTech, Beijing, Daxing, China